CLINICAL TRIAL: NCT04439032
Title: Multicenter Prospective Registry to Evaluate Use and Outcomes of NanoBone® Bone Graft Substitute in Spinal Fusion Surgery
Brief Title: Artoss Prospective Spine Registry Outcomes
Acronym: ASTRO
Status: Active, not recruiting | Type: Observational
Sponsor: Artoss Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SF-100
Record Dates: First submitted 2020-06-02; First posted 2020-06-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Spinal Fusion
Keywords: Bone Graft Substitute; Spinal Fusion; Degenerative Disc Disease; Scoliosis; Spine Deformity
MeSH Terms: conditions — Intervertebral Disc Degeneration; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spine Fusion using NanoBone: All patients in the study will be drawn from the individual surgeons' practice. Patients will be candidates for spinal fusion surgery after having failed conservative treatment or will have had spinal fusion surgery but have not completed their standard of care follow-up as determined by the surgeon's practice. In addition, the surgeon has determined that the use of a NanoBone product is or was clinically necessary for the patient.
  Interventions: Other: NanoBone Bone Graft Substitute

INTERVENTIONS:
Other: NanoBone Bone Graft Substitute — Synthetic, biodegradable bone grafting material that is composed of non-sintered nanocrystalline hydroxyapatite (HA) which is embedded in a silica gel matrix (amorphous SiO2). The ratio of HA/SiO2 has been chosen to optimize the rate of biodegradation for treatment of osseous defects in human bone. NanoBone does not contain any components of animal or human origin, eliminating the possibility of transmission of infection or disease.
  Other Names: nanoHA-SiO2

SUMMARY:
This prospective registry was designed as an observational study to ascertain how commercially available NanoBone Bone Graft is being used by surgeons performing spinal fusion as well as determining relevant patient outcomes.

DETAILED DESCRIPTION:
This multicenter prospective patient registry was developed with the aim of documenting how spine and neurosurgeons are utilizing the NanoBone products along with relevant patient outcomes. These outcomes include radiographic measures such as fusion outcome, instrumentation integrity, and clinical outcomes (symptom and function improvement) based on investigator and patient-based outcome assessments.

The primary objective of this study is to document and analyze the use of NanoBone products in spine fusion surgery (as a stand-alone bone graft, or in combination with local bone only, no other BGS or biologic product used) and determine both radiographic success and clinical outcomes. All product related adverse events will be documented, tabulated, and summarized.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient is diagnosed with a degenerative spine disorder requiring spinal fusion, has failed conservative treatment, and has decided to undergo surgery.
* The surgeon has determined that a NanoBone product is or was clinically indicated, and will use or have used the product as a stand-alone bone graft substitute or in combination with local autograft only (no iliac crest harvesting, other BGS, or biologic {defined as containing growth factors, cytokines, proteins, or cells} used).
* Patient capable of understanding the content of the Informed Consent Form
* Patient willing and able to participate in the registry protocol including SOC follow-up visits and clinical evaluations.
* Patient who has agreed to participate in the registry by providing consent according to the applicable local law and the Declaration of Helsinki.

Exclusion Criteria:• Severe vascular or neurological disease

* Uncontrolled diabetes
* Severe degenerative disease (other than degenerative disc disease)
* Severely impaired renal function
* Hypercalcemia, abnormal calcium metabolism
* Existing acute or chronic infections, especially at the site of the operation
* Inflammatory bone disease such as osteomyelitis
* Malignant tumors
* Patients who are or plan to become pregnant.
* Uncooperative patients who cannot or will not follow post-operative instruction, including individuals who abuse drugs and/or alcohol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients in the study will be drawn from the individual surgeons' practice. Patients will be candidates for spinal fusion surgery after having failed conservative treatment or will have had spinal fusion surgery but have not completed their standard of care follow-up as determined by the surgeon's practice. In addition, the surgeon has determined that the use of a NanoBone product is or was clinically necessary for the patient. The choice of a NanoBone product is or was independent of this research project. Only patients who have had NanoBone implanted and consent to participate and meet the inclusion-exclusion criteria will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success | 12-months
  Evidence of bony bridging between vertebral endplates and/or transverse processes of bone grafted vertebrae or absence of motion between vertebral bodies or both.

SECONDARY OUTCOMES:
Safety Evaluation | 12-months
  Occurrence of Complications or Adverse Events

OTHER OUTCOMES:
Clinical Success | 12-months
  Improvement from baseline in Visual Analog Scale (VAS) pain score (0= no pain, 10=worst possible pain)
Function | 12-months
  Improvement from baseline in Oswestry Disability Index (ODI) or Neck Disability Index (NDI) Scale (0=no disability-100=totally disabled)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cassidy, PhD, Study Director — Artoss Inc.
Locations (6):
- United States (6):
  - OrthoArizona, Chandler, Arizona
  - Sonoran Spine, Tempe, Arizona
  - SENTA Clinic, San Diego, California
  - Hartford Health Care, Hartford, Connecticut
  - OrthoBethesda, Bethesda, Maryland
  - Sam Shamsnia MD Neurosurgery, Biloxi, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://artossinc.com